CLINICAL TRIAL: NCT03882216
Title: Clinical Comparison of Pontic Site Development With Connective Tissue Graft Using Modified Pouch Technique Versus Pouch Technique: A Randomized Controlled Clinical Trial
Brief Title: Pontic Site Development With Connective Tissue Graft Using Modified Pouch Technique Versus Pouch Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Abdle Aziz Ammar, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5111987
Record Dates: First submitted 2019-02-14; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Ridge Deficency; Soft Tissue Augmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test group pouch technique (Experimental): free connective tissue graft augmentation using pouch technique
  Interventions: Procedure: soft tissue augmentation using pouch technique
- test group modified pouch technique (Experimental): free connective tissue graft augmentation using modified pouch technique
  Interventions: Procedure: soft tissue augmentation using modified pouch technique

INTERVENTIONS:
Procedure: soft tissue augmentation using pouch technique — crestal incision with split thickness flap without vertical releasing incision till the mucogingival line then apply the harvested connective tissue graft through it.
  Arms: test group pouch technique
Procedure: soft tissue augmentation using modified pouch technique — tunneling will be done at the pontic site till the mucogingival line then a distant vertical incision near the tunnel at the lining mucosa where the harvested connective tissue graft wll be applied .
  Arms: test group modified pouch technique

SUMMARY:
The study will be formed on two groups : the control group and the test group For both groups base line impressions will be taken before the surgery and a free gingival graft will be harvested from the palate and deepithelialized to obtain the free connective tissue graft then In the control group: the free connective tissue graft will be inserted through crestal pouch previously prepared using split thickness flap.

In the test group The free connective tissue graft will be slided through apical vertical incision in the pontic area previously tunneled.

Post operative casts will be obtained by taking impressions after three months and six months to evaluate the volumetric changes in the pontic area.

DETAILED DESCRIPTION:
Study settings: Study is to be conducted in the Oral Medicine and Periodontology department, Faculty of Dentistry - Cairo University, Egypt. Patients are to be selected from the outpatient clinic of the department of Oral Medicine and Periodontology-Cairo University Pre-surgical phase: Patients will be initially examined. All patients received oral hygiene instructions, and non-surgical periodontal treatment will be performed if necessary. At baseline, clinical periodontal measurements including plaque Index, bleeding on probing (BOP) , probing depth (PD) and clinical attachment level (CAL) will be recorded at teeth adjacent to the gap using a Williams's periodontal probe. Impressions will be taken using high viscosity impression material. Models will be cast in dental stone and used as the baseline reference for volumetric measurements. De-epithelialized connective tissue harvesting: The palatal sites will be anaesthetized with 0.3 ml of a solution of 4% Articaine and 0.001% Adrenalin. Graft harvesting will be performed by basic surgical techniques ). A rectangular shaped piece of mucosa will be harvested from the area of the hard palate by a split-thickness dissection. The graft will then be de-epithelialized, and the connective tissue graft will be used. Surgical site preparation for either control or intervention group: 1- Local anesthesia (2% lidocaine, 1: 100 000 epinephrine), incisions will be placed over the crest of the ridge reaching to alveolar bone. 2- Papillae will include in the incision line only when there is a loss of papillary height. 3- A deep supraperiosteal soft tissue pouch will be prepared by sharp dissection extending apically to the mucogingival line and to the neighboring teeth mesio-distally. 4- A rectangular shaped free gingival graft will be harvested from the contralateral palate using split thickness dissection.

Control group: -The graft will be de-epithelialized and the connective tissue graft will be inserted into the pouch that will be previously prepared at the recipient site and will be secured with two non-resorbable sutures at the labial and the palatal aspect. - Provisional restoration will be temporary cemented. -. Patient will be recalled after 14 days for suture removal.

Test group: Modified pouch technique -. De-epithelialization of the area that resembles in position and size the emergence profile of the pontic -. Tunnel preparation in the soft tissues buccal to the defect region using split thickness flap preparation. - Preparation of the pouch extends in a lateral direction to adjacent teeth and in an apical direction beyond the mucogingival line in order to ensure sufficient flap mobility. -. Flap preparation will also include elevation of the interproximal tissues lateral to the edentulous site. - Vertical releasing incision in the alveolar mucosa apical and distant to the defect will be done. -. The graft will be then drawn using positioning sutures. -. Provisional restoration will be temporary cemented on both abutments then double-crossed sutures are used for the fixation of the buccal soft-tissue complex, including the connective tissue graft. 8. Patient will be recalled after 14 days for suture removal. After the surgical volume augmentation procedure, clinical periodontal measurements will be recorded, impressions will be retaken and models will be cast at 3 and 6 months postoperative, In both control and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

1. Missing single tooth loss in anterior and premolar region.
2. Seibert Class I ridge defect.
3. Systemically free patients.
4. The healing period after the tooth extraction had to be at least 3 months prior to the surgical procedures.

Exclusion Criteria:

1. Smokers
2. Occlusal trauma at site of graft
3. Pregnancy and lactation
4. Severe gagging reflex

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-20 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
volumetric changes at the pontic site | 6 months
  To evaluate the volumetric changes between the baseline and 6 months postoperatively all the cast stone models will be digitized using lab based optical scannerDigital cast models will be reproduced resembling different time points during treatmentSuperimposing the different models of the same case using the best fit algorithm by taking the tooth surfaces as references The area of pontic site will be defined by the mesial and distal papillary midline, the mucogingival line, and the alveolar crest So any volumetric changes between digitalized superimposed casts can be measured.

SECONDARY OUTCOMES:
Postoperative pain - through Visual Analogue Scale | 14 days
  Pain score reported by the patient directly through Visual Analogue Scale score (between 0 and 10. 0: no pain, 1: minimal pain, 5:moderate pain, 10: severe pain) VAS will be recorded at day 14